CLINICAL TRIAL: NCT01892436
Title: A Three-year Extension Study to Evaluate the Long Term Efficacy, Safety and Tolerability of Secukinumab in Patients With Active Psoriatic Arthritis
Brief Title: Extension Study up to 3 Years for Secukinumab in Psoriatic Arthritis
Acronym: FUTURE 1 ext
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAIN457F2306E1; 2013-001241-13 (EudraCT Number)
Record Dates: First submitted 2013-07-01; First posted 2013-07-04 (Estimated); Results first posted 2019-06-12 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-05

CONDITIONS: Psoriatic Arthritis
Keywords: Extension study, psoriatic arthritis, pre-filled syringe
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Secukinumab 75mg (Experimental): Subjects continued to receive secukinumab 75mg in PFS (same dose as that was received in core study CAIN457F2306) every 4 weeks up to Week 256. From Week 156, patients may have been escalated to 150 mg or 300 mg as judged appropriate by investigator
  Interventions: Drug: Secukinumab
- Secukinumab 150mg (Experimental): Subjects continued to receive secukinumab 150mg in PFS (same dose as that was received in core study CAIN457F2306) every 4 weeks up to Week 256. From Week 156, patients may have been escalated to 300 mg as judged appropriate by the investigator
  Interventions: Drug: Secukinumab
- Placebo - AIN457A 75mg (Experimental): Placebo (for maintaining the blind till Week 152): Placebo to secukinumab 0.5 mL solution solution for injection was provided in PFS for s.c. administration (a single use pre-filled 1mL long glass syringe). It contained a mixture of inactive excipients, matching the composition of secukinumab 75mg
  Interventions: Drug: Secukinumab; Drug: Placebo
- Placebo - AIN457 150mg (Experimental): Placebo (for maintaining the blind till Week 152): Placebo to secukinumab 1 mL solution for injection was provided in PFS for s.c. administration (a single use pre-filled 1mL long glass syringe). It contained a mixture of inactive excipients, matching the composition of secukinumab 150 mg
  Interventions: Drug: Secukinumab; Drug: Placebo

INTERVENTIONS:
Drug: Secukinumab — Secukinumab is a human monoclonal antibody. Monoclonal antibodies are proteins that recognize and bind to unique proteins that your body produces. Secukinumab binds and reduces the activity of a cytokine (a "messenger" protein in the body) called Interleukin 17 (IL-17).
  Other Names: AIN457
Drug: Placebo — Placebo
  Other Names: Placebo - AIN457A
  Arms: Placebo - AIN457 150mg; Placebo - AIN457A 75mg

SUMMARY:
This study was designed as a 3-year extension to the phase III core study CAIN457F2306. It aimed to provide continuous treatment with secukinumab in pre-filled syringes (PFS) for subjects who completed the core study CAIN457F2306, to obtain further long term efficacy, safety and tolerability information in subjects with active psoriatic arthritis receiving secukinumab every 4 weeks. At Week 104 of the study CAIN457F2306, eligible subjects completed the assessments associated with the core study visit and subsequently continued in this extension study on the same dose that they were receiving during the core study. The regular assessments of disease activity ensure that subjects who are experienced worsening of disease in any of the treatment groups could exit the study upon their own wish or based on the advice of the investigator at any time.

ELIGIBILITY:
Inclusion criteria

* Subjects must be able to understand and communicate with the investigator and comply with the requirements of the study and must give a written, signed and dated informed consent before any study assessment is performed
* Subjects must have participated in core study CAIN457F2306, and must have completed the entire treatment period
* Subjects must be deemed by the investigator to benefit from continued secukinumab therapy

Exclusion criteria

* Any subject taking other concomitant biologic immunomodulating agent(s) except secukinumab
* Any subject who is deemed not to be benefiting from the study treatment based upon lack of improvement or worsening of their symptoms
* Pregnant or nursing (lactating) women
* Women of child-bearing potential, unless they are using effective methods of contraception during the entire study or longer if required by locally approved prescribing information (e.g., 20 weeks in EU)

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2013-09-30 (Actual); Primary Completion 2018-01-11 (Actual); Study Completion 2018-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (84):
- United States (21):
  - Novartis Investigative Site, Anniston, Alabama
  - Novartis Investigative Site, Mesa, Arizona
  - Novartis Investigative Site, Paradise Valley, Arizona
  - Novartis Investigative Site, Upland, California
  - Novartis Investigative Site, Tamarac, Florida
  - Novartis Investigative Site, Eagan, Minnesota
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Freehold, New Jersey
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Duncansville, Pennsylvania
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Columbia, South Carolina
  - Novartis Investigative Site, Jackson, Tennessee
  - Novartis Investigative Site, Benbrook, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, League City, Texas
  - Novartis Investigative Site, Mesquite, Texas
  - Novartis Investigative Site, Seattle, Washington
- Argentina (5):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, CABA
  - Novartis Investigative Site, Córdoba
- Australia (2):
  - Novartis Investigative Site, Maroochydore, Queensland
  - Novartis Investigative Site, Malvern East, Victoria
- Belgium (3):
  - Novartis Investigative Site, Genk
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Leuven
- Brazil (2):
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, São Paulo, São Paulo
- Bulgaria (3):
  - Novartis Investigative Site, Sevlievo, Gabrovo
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Sofia
- Canada (4):
  - Novartis Investigative Site, St. John's, Newfoundland and Labrador
  - Novartis Investigative Site, Newmarket, Ontario
  - Novartis Investigative Site, Waterloo, Ontario
  - Novartis Investigative Site, Trois-Rivières, Quebec
- Czechia (3):
  - Novartis Investigative Site, Bruntál, Czech Republic
  - Novartis Investigative Site, Uherské Hradiště, Czech Republic
  - Novartis Investigative Site, Zlín, Czech Republic
- Germany (10):
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Gommern
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hildesheim
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Ratingen
  - Novartis Investigative Site, Zerbst
- Israel (4):
  - Novartis Investigative Site, Ashkelon
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Italy (4):
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Prato, PO
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Verona, VR
- Philippines (6):
  - Novartis Investigative Site, Lipa City, Batangas
  - Novartis Investigative Site, Dasmariñas, Cavite
  - Novartis Investigative Site, Manila, National Capital Region
  - Novartis Investigative Site, Las Piñas
  - Novartis Investigative Site, Manila
  - Novartis Investigative Site, Quezon City
- Poland (2):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Warsaw
- Russia (5):
  - Novartis Investigative Site, Kemerovo
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Yaroslavl
  - Novartis Investigative Site, Yekaterinburg
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Lučenec, Slovakia
- Thailand (3):
  - Novartis Investigative Site, Khon Kaen, THA
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
- United Kingdom (5):
  - Novartis Investigative Site, Leytonstone, London
  - Novartis Investigative Site, Cannock, Staffordshire
  - Novartis Investigative Site, Bradford, West Yorkshire
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Mease PJ, Kavanaugh A, Reimold A, Tahir H, Rech J, Hall S, Geusens P, Pellet P, Delicha EM, Mpofu S, Pricop L. Secukinumab in the treatment of psoriatic arthritis: efficacy and safety results through 3 years from the year 1 extension of the randomised phase III FUTURE 1 trial. RMD Open. 2018 Aug 13;4(2):e000723. doi: 10.1136/rmdopen-2018-000723. eCollection 2018. PMID 30167329

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The extension FAS (N=457) comprised all patients enrolled in the extension with at least 1 post baseline efficacy assessment during the extension study. 3 patients signed the ICF but had no efficacy assessments during the extension study and were not included in extension FAS.
Pre-assignment Details: Of the 457 patients in the extension FAS, 380 (83.2%) completed 260 weeks of treatment (84.4% in the secukinumab 10 mg/kg-75 mg group, 82.0% in the secukinumab 10 mg/kg-150 mg group, 85.1% in the placebo-secukinumab 75 mg group and 81.3% in the placebo-secukinumab 150 mg group)
Groups:
- Placebo - AIN457A 75mg: Placebo (for maintaining the blind till Week 152): Placebo to secukinumab 1.0 mL solution for injection was provided in PFS for s.c. administration (a single use pre-filled 1mL long glass syringe). It contained a mixture of inactive excipients, matching the composition of secukinumab 75mg. Participants also received secukinumab 75mg from week 16/24. Patients may have been escalated to 150 mg or 300 mg as judged appropriate by investigator
- Placebo - AIN457 150mg: Placebo (for maintaining the blind till Week 152): Placebo to secukinumab 0.5mL solution for injection was provided in PFS for s.c. administration (a single use pre-filled 1mL long glass syringe). It contained a mixture of inactive excipients, matching the composition of secukinumab 150 mg. Participants also received secukinumab 150 mg from week 16/24. patients may have been escalated to 300mg or 300 mg as judged appropriate by investigator
Period: Overall Study
Arm/Group | Secukinumab 75mg | Secukinumab 150mg | Placebo - AIN457A 75mg | Placebo - AIN457 150mg
Started | 147 | 161 | 74 | 75
Completed | 124 | 132 | 63 | 61
Not Completed | 23 | 29 | 11 | 14
Not completed — Withdrawal by Subject | 8 | 15 | 4 | 4
Not completed — Death | 1 | 1 | 0 | 0
Not completed — Physician Decision | 2 | 1 | 0 | 1
Not completed — Pregnancy | 0 | 2 | 1 | 0
Not completed — Technical problems | 2 | 1 | 1 | 1
Not completed — Lack of Efficacy | 1 | 2 | 2 | 2
Not completed — Lost to Follow-up | 1 | 1 | 1 | 3
Not completed — non-compliance with treatment | 1 | 0 | 0 | 0
Not completed — Adverse Event | 7 | 6 | 2 | 3

BASELINE CHARACTERISTICS:
Population: Extension Full Analysis Set (extension FAS) is comprised all patients enrolled in the extension study who had at least one post baseline assessment of efficacy during the extension period. Patients were analyzed according to the treatment they were assigned.
Groups:
- Secukinumab 75mg: Subjects initially continued to receive secukinumab 75mg in PFS (same dose as that was received in core study CAIN457F2306) every 4 weeks up to Week 256. From Week 156, patients may have been escalated to 150 mg or 300 mg as judged appropriate by investigator
- Total: Total of all reporting groups
Arm/Group | Secukinumab 75mg | Secukinumab 150mg | Placebo - AIN457A 75mg | Placebo - AIN457 150mg | Total
Number analyzed (Participants) | 147 | 161 | 74 | 75 | 457
Age, Customized [Number; unit: Count of Participants] — Age groups are reported cumulatively so categories are not mutually exclusive.
  Count of Participants
    <65 | 132 | 145 | 72 | 71 | 420
    >=65 | 15 | 16 | 2 | 4 | 37
    >=75 | 1 | 0 | 1 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 83 | 40 | 38 | 242
  Male | 66 | 78 | 34 | 37 | 215
Race/Ethnicity, Customized [Number; unit: Count of participants]
  White | 118 | 130 | 51 | 58 | 357
  Black or African American | 1 | 1 | 0 | 0 | 2
  Asian | 27 | 29 | 23 | 16 | 95
  Other | 1 | 1 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subject Who Reached (American College of Rheumatology Score of 20) ACR20
Description: Proportion of subjects with a positive clinical response to treatment (individual improvement) in disease activity according to ACR20 criteria if he/she has at least 20% improvement in 1. Tender 68-joint count 2. Swollen 66-joint count and 3. At least 3 of the following 5 measures:
  * Patient's assessment of Psoriatic Arthritis (PsA) pain
  * Patient's global assessment of disease activity
  * Physician's global assessment of disease activity
  * Subject self-assessed disability (Health-Assessment Questionnaire [HAQ-DI] score)
  * Acute phase reactant (hsCRP or ESR)
Time Frame: weeks 116, 128, 140, 156, 180, 208, 232 and 260
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Secukinumab 75mg | Secukinumab 150mg | Placebo - AIN457A 75mg | Placebo - AIN457 150mg
Number analyzed (Participants) | 147 | 161 | 74 | 75
percentage of participants
  week 116 | 71.3 [63.1 to 78.4] | 73.9 [66.0 to 80.5] | 73.2 [61.2 to 82.7] | 73.6 [61.7 to 83.0]
  week 128 | 69.7 [61.4 to 77.0] | 72.9 [65.1 to 79.6] | 76.8 [64.8 to 85.8] | 74.6 [62.7 to 83.9]
  week 140 | 69.8 [61.3 to 77.1] | 71.1 [63.1 to 78.0] | 79.2 [67.7 to 87.5] | 69.4 [57.3 to 79.5]
  week 156 | 64.3 [55.8 to 72.0] | 76.1 [68.5 to 82.4] | 75.3 [63.6 to 84.4] | 67.6 [55.6 to 77.7]
  week 180 | 73.0 [64.6 to 80.0] | 72.5 [64.1 to 79.6] | 74.6 [62.3 to 84.1] | 67.7 [54.8 to 78.5]
  week 208 | 72.8 [64.4 to 79.9] | 66.9 [58.5 to 74.3] | 75.0 [62.8 to 84.4] | 68.2 [55.4 to 78.8]
  week 232 | 79.5 [71.3 to 86.0] | 69.5 [60.7 to 77.0] | 83.3 [71.7 to 91.0] | 80.3 [67.8 to 89.0]
  week 260 | 77.2 [68.7 to 83.9] | 67.9 [59.1 to 75.7] | 78.8 [66.7 to 87.5] | 77.4 [64.7 to 86.7]

2. Primary Outcome: Proportion of Subjects Who Reached ACR50
Description: Proportion of subjects that have a positive clinical response to treatment (individual improvement) in disease activity according to ACR50 criteria if he/she has at least 50% improvement in 1. Tender 68-joint count 2. Swollen 66-joint count and 3. At least 3 of the following 5 measures:
  * Patient's assessment of PsA pain
  * Patient's global assessment of disease activity
  * Physician's global assessment of disease activity
  * Subject self-assessed disability (Health-Assessment Questionnaire [HAQ-DI] score)
  * Acute phase reactant (hsCRP or ESR)
Time Frame: weeks 116, 128, 140, 156, 180, 208, 232 and 260
Population: Extension FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Secukinumab 75mg | Secukinumab 150mg | Placebo - AIN457A 75mg | Placebo - AIN457 150mg
Number analyzed (Participants) | 147 | 161 | 74 | 75
percentage of participants
  week 116 | 43.4 [35.2 to 51.9] | 51.0 [42.8 to 59.1] | 49.3 [37.3 to 61.3] | 47.2 [35.5 to 59.3]
  week 128 | 43.7 [35.4 to 52.2] | 52.9 [44.8 to 60.9] | 56.5 [44.1 to 68.2] | 53.5 [41.4 to 65.3]
  week 140 | 41.7 [33.5 to 50.4] | 48.7 [40.5 to 56.9] | 51.4 [39.4 to 63.2] | 44.4 [32.9 to 56.6]
  week 156 | 39.2 [31.2 to 47.7] | 56.1 [47.9 to 64.0] | 52.1 [40.1 to 63.8] | 47.3 [35.7 to 59.2]
  week 180 | 43.1 [34.7 to 51.8] | 45.7 [37.2 to 54.3] | 52.2 [39.8 to 64.4] | 50.8 [38.2 to 63.3]
  week 208 | 44.9 [36.4 to 53.6] | 46.9 [38.6 to 55.3] | 52.9 [40.5 to 65.0] | 53.0 [40.4 to 65.3]
  week 232 | 49.6 [40.7 to 58.6] | 53.4 [44.5 to 62.1] | 53.0 [40.4 to 65.3] | 50.8 [37.8 to 63.7]
  week 260 | 51.2 [42.2 to 60.1] | 52.7 [43.8 to 61.4] | 60.6 [47.8 to 72.2] | 50.0 [37.2 to 62.8]

3. Primary Outcome: Proportion of Subjects Who Reached ACR70
Description: Proportion of subjects that have a positive clinical response to treatment (individual improvement) in disease activity according to ACR70 criteria if he/she has at least 70% improvement in 1. Tender 68-joint count 2. Swollen 66-joint count and 3. At least 3 of the following 5 measures:- Patient's assessment of PsA pain
  * Patient's global assessment of disease activity
  * Physician's global assessment of disease activity
  * Subject self-assessed disability (Health-Assessment Questionnaire [HAQ-DI] score)
  * Acute phase reactant (hsCRP or ESR)
Time Frame: weeks 116, 128, 140, 156, 180, 208, 232 and 260
Population: Extension FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Secukinumab 75mg | Secukinumab 150mg | Placebo - AIN457A 75mg | Placebo - AIN457 150mg
Number analyzed (Participants) | 147 | 161 | 74 | 75
percentage of participants
  week 116 | 23.8 [17.2 to 31.8] | 30.1 [23.1 to 38.1] | 28.2 [18.4 to 40.3] | 29.2 [19.3 to 41.2]
  week 128 | 24.6 [18.0 to 32.7] | 31.0 [23.9 to 39.0] | 34.8 [24.0 to 47.3] | 23.9 [14.9 to 35.8]
  week 140 | 27.3 [20.3 to 35.7] | 28.3 [21.4 to 36.3] | 33.3 [22.9 to 45.5] | 27.8 [18.2 to 39.8]
  week 156 | 25.9 [19.1 to 34.0] | 32.9 [25.7 to 41.0] | 26.0 [16.8 to 37.8] | 27.0 [17.7 to 38.8]
  week 180 | 27.0 [20.0 to 35.4] | 31.2 [23.7 to 39.7] | 31.3 [20.9 to 44.0] | 27.7 [17.7 to 40.4]
  week 208 | 25.7 [18.8 to 34.1] | 31.0 [23.8 to 39.3] | 32.4 [21.8 to 44.9] | 28.8 [18.6 to 41.4]
  week 232 | 35.4 [27.3 to 44.5] | 32.1 [24.3 to 40.9] | 37.9 [26.5 to 50.7] | 34.4 [23.0 to 47.8]
  week 260 | 33.9 [25.9 to 42.9] | 37.4 [29.2 to 46.3] | 37.9 [26.5 to 50.7] | 33.9 [22.6 to 47.1]

4. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI)
Description: Changes from baseline in score of the disability assessment component of the HAQ (Health Assessment Questionnaire - Disability Index). The HAQ-DI, assesses a subject's level of functional ability and includes questions of fine movements of the upper extremity, locomotor activities of the lower extremity, and activities that involve both upper and lower extremities.
  Health Assessment Questionnaire - Disability Index (HAQ-DI) ranges from 0 (no disability) to 3 (very severe disability)
Time Frame: weeks 116, 128, 140, 156, 180, 208, 232 and 260
Population: Extension FAS
Measure: Mean (Standard Deviation); unit: change in scores
Arm/Group | Secukinumab 75mg | Secukinumab 150mg | Placebo - AIN457A 75mg | Placebo - AIN457 150mg
Number analyzed (Participants) | 147 | 161 | 74 | 75
change in scores
  week 116 | -0.4537 (0.60617) | -0.4592 (0.56155) | -0.5642 (0.56722) | -0.4115 (0.66721)
  week 128 | -0.4171 (0.61192) | -0.4619 (0.55835) | -0.5143 (0.55599) | -0.3750 (0.69661)
  week 140 | -0.4448 (0.61406) | -0.4713 (0.58791) | -0.4635 (0.56037) | -0.3507 (0.69221)
  week 156 | -0.4236 (0.61896) | -0.4266 (0.57491) | -0.5068 (0.62548) | -0.3159 (0.73507)
  week 180 | -0.4617 (0.61472) | -0.4305 (0.59901) | -0.5698 (0.65258) | -0.3538 (0.71246)
  week 208 | -0.4463 (0.57130) | -0.3857 (0.59304) | -0.5531 (0.62622) | -0.3447 (0.74745)
  week 232 | -0.4710 (0.60931) | -0.4122 (0.60461) | -0.5777 (0.66930) | -0.3952 (0.72115)
  week 260 | -0.4821 (0.61170) | -0.4036 (0.58334) | -0.5038 (0.61039) | -0.3730 (0.71306)

5. Secondary Outcome: Minimal Clinically Important Difference (MCID) in Health Assessment Questionnaire Disability Index (HAQ-DI)
Description: Percentage of subjects with improvements from baseline in HAQ-DI meeting or exceeding minimal clinically important difference (MCID=0.3). The HAQ-DI, assesses a subject's level of functional ability and includes questions of fine movements of the upper extremity, locomotor activities of the lower extremity, and activities that involve both upper and lower extremities.
Time Frame: weeks 116, 128, 140, 156, 180, 208, 232 and 260
Population: Extension FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Secukinumab 75mg | Secukinumab 150mg | Placebo - AIN457A 75mg | Placebo - AIN457 150mg
Number analyzed (Participants) | 147 | 161 | 74 | 75
percentage of participants
  week 116 | 53.1 [44.6 to 61.5] | 52.3 [44.1 to 60.4] | 63.9 [51.7 to 74.6] | 50.0 [38.1 to 61.9]
  week 128 | 52.8 [44.3 to 61.2] | 51.9 [43.8 to 60.0] | 57.1 [44.8 to 68.7] | 54.9 [42.7 to 66.6]
  week 140 | 55.4 [46.7 to 63.7] | 52.3 [44.1 to 60.4] | 56.9 [44.8 to 68.4] | 48.6 [36.8 to 60.6]
  week 156 | 52.8 [44.3 to 61.1] | 52.3 [44.1 to 60.3] | 60.8 [48.7 to 71.7] | 44.6 [33.2 to 56.6]
  week 180 | 56.9 [48.2 to 65.3] | 51.5 [42.8 to 60.1] | 61.2 [48.5 to 72.6] | 47.7 [35.3 to 60.4]
  week 208 | 53.3 [44.6 to 61.9] | 50.0 [41.6 to 58.4] | 59.4 [46.9 to 70.9] | 48.5 [36.1 to 61.0]
  week 232 | 55.2 [46.1 to 64.0] | 48.9 [40.1 to 57.7] | 59.1 [46.3 to 70.8] | 52.5 [39.4 to 65.2]
  week 260 | 55.6 [46.5 to 64.3] | 48.9 [40.1 to 57.7] | 59.1 [46.3 to 70.8] | 53.2 [40.2 to 65.8]

6. Secondary Outcome: Change From Baseline in Disease Activity Score-CRP (DAS28)
Description: Changes in DAS28 (utilizing hsCRP) from baseline up to Month 60. The DAS28 is a measure of disease activity in PsA based on Swollen and Tender Joint Counts (out of a total of 28), hsCRP and the Patient's Global Assessment of Disease Activity. A DAS28 score greater than 5.1 implies active disease, equal to or less than 3.2 low disease activity, and less than 2.6 remission. This measure represents change in scores - not the actual scores.
  DAS28 is a combined measure of disease activity based on the following formula:
  DAS28-CRP = 0.56*TJC28^0.5 + 0.28*SJC28^0.5 + 0.36*ln(CRP+1) + 0.014*PGA + 0.96 The greater the score is, the more the disease activity exists. Remission is defined as DAS28-CRP < 2.6 Low disease activity is defined as DAS28-CRP < 3.2 The minimum value can be 0.96 (not applicable in our study due to the inclusion/exclusion criteria regarding tender, swollen joints). There is no maximum expected value for this score
Time Frame: weeks 116, 128, 140, 156, 180, 208, 232 and 260
Population: Extension FAS
Measure: Mean (Standard Deviation); unit: change in scores
Arm/Group | Secukinumab 75mg | Secukinumab 150mg | Placebo - AIN457A 75mg | Placebo - AIN457 150mg
Number analyzed (Participants) | 147 | 161 | 74 | 75
change in scores
  week 116 | -2.044 (1.3382) | -1.904 (1.3165) | -2.282 (1.2732) | -1.853 (1.2737)
  week 128 | -2.013 (1.3446) | -1.962 (1.2900) | -2.333 (1.2815) | -2.031 (1.3290)
  week 140 | -2.074 (1.3224) | -1.912 (1.2246) | -2.412 (1.3059) | -1.830 (1.3136)
  week 156 | -1.844 (1.4923) | -1.942 (1.3195) | -2.109 (1.3188) | -1.743 (1.3630)
  week 180 | -2.058 (1.3760) | -1.937 (1.2674) | -2.327 (1.2339) | -1.867 (1.4590)
  week 208 | -2.042 (1.2907) | -1.767 (1.4574) | -2.344 (1.3351) | -1.862 (1.4708)
  week 232 | -2.225 (1.2570) | -2.046 (1.2590) | -2.611 (1.3247) | -2.286 (1.2102)
  week 260 | -2.112 (1.2664) | -2.074 (1.3146) | -2.506 (1.3774) | -2.099 (1.2466)

7. Secondary Outcome: Percentage of Subjects Achieving Low Disease Activity
Description: Percentage of subjects achieving low disease activity (DAS28 ≤ 3.2). The DAS28 is a measure of disease activity in PsA based on Swollen and Tender Joint Counts (out of a total of 28), hsCRP and the Patient's Global Assessment of Disease Activity. A DAS28 score greater than 5.1 implies active disease, equal to or less than 3.2 low disease activity, and less than 2.6 remission
Time Frame: weeks 116, 128, 140, 156, 180, 208, 232 and 260
Population: Extension FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Secukinumab 75mg | Secukinumab 150mg | Placebo - AIN457A 75mg | Placebo - AIN457 150mg
Number analyzed (Participants) | 147 | 161 | 74 | 75
percentage of participants
  week 116 | 70.3 [62.1 to 77.5] | 64.7 [56.5 to 72.1] | 70.4 [58.2 to 80.4] | 63.9 [51.7 to 74.6]
  week 128 | 69.5 [61.1 to 76.8] | 69.9 [61.9 to 76.8] | 75.4 [63.3 to 84.6] | 68.6 [56.2 to 78.9]
  week 140 | 72.9 [64.6 to 79.9] | 66.0 [57.8 to 73.4] | 75.0 [63.2 to 84.1] | 65.3 [53.1 to 75.9]
  week 156 | 63.4 [54.8 to 71.2] | 67.9 [59.9 to 75.1] | 61.6 [49.5 to 72.6] | 58.9 [46.8 to 70.1]
  week 180 | 71.2 [62.8 to 78.4] | 70.1 [61.6 to 77.4] | 65.7 [53.0 to 76.6] | 68.8 [55.8 to 79.4]
  week 208 | 71.7 [63.3 to 78.9] | 65.8 [57.4 to 73.3] | 67.2 [54.5 to 77.9] | 71.2 [58.6 to 81.4]
  week 232 | 75.2 [66.7 to 82.2] | 73.5 [65.0 to 80.6] | 79.4 [67.0 to 88.1] | 84.7 [72.5 to 92.4]
  week 260 | 74.4 [65.8 to 81.5] | 75.0 [66.6 to 81.9] | 76.9 [64.5 to 86.1] | 77.4 [64.7 to 86.7]

8. Secondary Outcome: Percentage of Subjects Achieving Disease Remission (DAS28<2.6)
Description: Percentage of subjects achieving disease remission (DAS28<2.6). The DAS28 is a measure of disease activity in PsA based on Swollen and Tender Joint Counts (out of a total of 28), hsCRP and the Patient's Global Assessment of Disease Activity. A DAS28 score greater than 5.1 implies active disease, equal to or less than 3.2 low disease activity, and less than 2.6 remission
Time Frame: weeks 116, 128, 140, 156, 180, 208, 232 and 260
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Secukinumab 75mg | Secukinumab 150mg | Placebo - AIN457A 75mg | Placebo - AIN457 150mg
Number analyzed (Participants) | 147 | 161 | 74 | 75
percentage of participants
  week 116 | 52.4 [44.0 to 60.7] | 50.3 [42.2 to 58.5] | 47.9 [36.0 to 60.0] | 45.8 [34.2 to 57.9]
  week 128 | 54.6 [46.0 to 62.9] | 49.4 [41.3 to 57.4] | 55.1 [42.7 to 66.9] | 57.1 [44.8 to 68.7]
  week 140 | 58.6 [49.9 to 66.7] | 46.7 [38.5 to 55.0] | 55.6 [43.4 to 67.1] | 51.4 [39.4 to 63.2]
  week 156 | 48.6 [40.2 to 57.1] | 52.6 [44.4 to 60.6] | 43.8 [32.4 to 55.9] | 46.6 [35.0 to 58.6]
  week 180 | 54.7 [46.0 to 63.1] | 53.3 [44.6 to 61.8] | 49.3 [37.0 to 61.6] | 58.6 [46.2 to 70.0]
  week 208 | 56.5 [47.8 to 64.8] | 52.1 [43.7 to 60.3] | 55.2 [42.6 to 67.2] | 53.0 [40.4 to 65.3]
  week 232 | 64.3 [55.4 to 72.4] | 61.4 [52.5 to 69.6] | 65.1 [51.9 to 76.4] | 69.5 [56.0 to 80.5]
  week 260 | 55.0 [46.0 to 63.7] | 58.3 [49.4 to 66.7] | 64.6 [51.7 to 75.8] | 66.1 [52.9 to 77.4]

ADVERSE EVENTS:
Time Frame: week 260
Description: Safety analysis is based on the actual dose received. Pts who escalated from 75mg to 150mg or 300mg are also analyzed at the escalated dose Any AIN75: 202 AIN75 + 93 PBO-AIN150 - 3 PBO-AIN150 (re-randomized but not exposed) = 292 Any AIN150: 202 AIN150 + 94 PBO-AIN150 + 178 Up-titrators from 75mg -1 PBO-AIN150 (re-randomized but not exposed) = 473 Any 300: 165 Up-titrators Placebo: 149 pts entered the extension and were on PBO up to wks 16/24. Also, add 53 PBOs who did not enter the extension
Groups:
- Any AIN457 75 mg: Any AIN457 75 mg
- Any AIN457 150 mg: Any AIN457 150 mg
- Any AIN457 300 mg: Any AIN457 300 mg
Arm/Group | Any AIN457 75 mg | Any AIN457 150 mg | Any AIN457 300 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 3/292 | 3/473 | 0/165 | 0/202
Serious Adverse Events (participants affected / at risk) | 48/292 | 96/473 | 10/165 | 11/202
Other Adverse Events (participants affected / at risk) | 197/292 | 264/473 | 47/165 | 63/202
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Any AIN457 75 mg (N=292) | Any AIN457 150 mg (N=473) | Any AIN457 300 mg (N=165) | Placebo (N=202)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 2 | 0 | 0
Angina pectoris (Cardiac disorders) | 2 | 2 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 1 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 2 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 2 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 2 | 0 | 1
Coronary artery insufficiency (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 3 | 0 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 2 | 0 | 0 | 0
Basedow's disease (Endocrine disorders) | 0 | 1 | 0 | 0
Goitre (Endocrine disorders) | 2 | 0 | 0 | 0
Ocular myasthenia (Eye disorders) | 1 | 0 | 0 | 0
Abdominal adhesions (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Femoral hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Impaired healing (General disorders) | 0 | 2 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 4 | 0 | 1
Peripheral swelling (General disorders) | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 2 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Chronic hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Abdominal sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 0
Appendiceal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 2 | 4 | 0 | 0
Dengue fever (Infections and infestations) | 1 | 0 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 3 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 1 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Intervertebral discitis (Infections and infestations) | 0 | 1 | 0 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Lung abscess (Infections and infestations) | 0 | 1 | 0 | 0
Necrotising fasciitis (Infections and infestations) | 1 | 0 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 4 | 1 | 0
Post procedural infection (Infections and infestations) | 0 | 1 | 0 | 0
Prostatitis Escherichia coli (Infections and infestations) | 1 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 1 | 0 | 0 | 0
Salpingo-oophoritis (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 2 | 0 | 0 | 0
Septic shock (Infections and infestations) | 2 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Streptococcal infection (Infections and infestations) | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0
Typhoid fever (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 2 | 1 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0
Wound infection staphylococcal (Infections and infestations) | 0 | 1 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Eyelid injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Periprosthetic osteolysis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Traumatic liver injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Limb asymmetry (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 7 | 1 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 5 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Intraductal papilloma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Laryngeal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Pleomorphic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 0
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Squamous cell carcinoma of pharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Hemiplegia (Nervous system disorders) | 1 | 0 | 0 | 0
Intracranial venous sinus thrombosis (Nervous system disorders) | 1 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Thrombotic stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 2 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 2 | 0 | 0
Adenomyosis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Adnexa uteri cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Pelvic adhesions (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 1
Pelvic venous thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Polyarteritis nodosa (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Any AIN457 75 mg (N=292) | Any AIN457 150 mg (N=473) | Any AIN457 300 mg (N=165) | Placebo (N=202)
Diarrhoea (Gastrointestinal disorders) | 23 | 38 | 1 | 6
Nausea (Gastrointestinal disorders) | 17 | 14 | 3 | 2
Vomiting (Gastrointestinal disorders) | 15 | 8 | 0 | 1
Bronchitis (Infections and infestations) | 24 | 35 | 9 | 6
Gastroenteritis (Infections and infestations) | 10 | 30 | 2 | 2
Nasopharyngitis (Infections and infestations) | 70 | 101 | 14 | 11
Pharyngitis (Infections and infestations) | 15 | 22 | 0 | 0
Sinusitis (Infections and infestations) | 17 | 26 | 3 | 4
Upper respiratory tract infection (Infections and infestations) | 62 | 91 | 10 | 12
Urinary tract infection (Infections and infestations) | 21 | 27 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 | 30 | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 30 | 33 | 3 | 2
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 23 | 27 | 2 | 2
Headache (Nervous system disorders) | 31 | 42 | 1 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 30 | 3 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 20 | 19 | 1 | 4
Psoriasis (Skin and subcutaneous tissue disorders) | 23 | 23 | 2 | 1
Hypertension (Vascular disorders) | 27 | 33 | 7 | 5

LIMITATIONS AND CAVEATS:
Observed data is reported for outcome measures

The non-fatal adverse events are reported under "Serious Adverse Events"

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-07-22): https://cdn.clinicaltrials.gov/large-docs/36/NCT01892436/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-12): https://cdn.clinicaltrials.gov/large-docs/36/NCT01892436/SAP_001.pdf